CLINICAL TRIAL: NCT00443976
Title: A Phase I Study of AT9283 Given As a 24 Hour Infusion on Days 1 and 8 Every Three Weeks in Patients With Advanced Incurable Malignancy
Brief Title: Aurora Kinase Inhibitor AT9283 in Treating Patients With Advanced or Metastatic Solid Tumors or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I181; CDR0000523837 (Registry Identifier: PDQ); CAN-NCIC-IND181 (Registry Identifier: NCI US - Physician Data Query); ASTEX-CAN-NCIC-IND181 (Registry Identifier: Astex Therapeutics Inc.)
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Non-Hodgkins Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 2 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; recurrent adult grade III lymphomatoid granulomatosis; adult grade III lymphomatoid granulomatosis; Waldenstrom macroglobulinemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AT9283 (Experimental)
  Interventions: Drug: Aurora kinase inhibitor AT9283

INTERVENTIONS:
Drug: Aurora kinase inhibitor AT9283 — The starting dose of AT9283 will be 1.5 mg/m2 given as a 24 hour IV infusion on Days 1 and 8 every three weeks.

SUMMARY:
RATIONALE: Aurora kinase inhibitor AT9283 (AT9283) may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of AT9283 in treating patients with advanced or metastatic solid tumors or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of Aurora kinase inhibitor AT9283 (AT9283) in patients with incurable advanced or metastatic solid tumors or non-Hodgkin's lymphoma.
* Determine the safety, tolerability, toxicity profile, dose-limiting toxicity, and pharmacokinetic profile of this drug in these patients.
* Correlate the toxicity profile with the pharmacokinetics of this drug in these patients.
* Assess, preliminarily, evidence of antitumor activity of this drug in these patients.
* Determine the pharmacodynamic activity of this drug in these patients and correlate with biological endpoints.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive Aurora kinase inhibitor AT9283 (AT9283) IV over 24 hours on days 1 and 8 . Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of AT9283 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. The dose preceding the MTD is the recommended phase II dose (RPTD). Up to 8 additional patients are treated at the RPTD.

Patients treated at the RPTD undergo skin and tumor tissue biopsy and blood collection at baseline and on days 2 and/or 3. Samples are examined by pharmacokinetic and pharmacodynamic analysis, including immunohistochemistry, immunocytochemistry, western blotting, immunoenzyme techniques, flow cytometry, and reverse transcriptase-polymerase chain reaction, for biological markers.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months until disease progression.

PROJECTED ACCRUAL: Up to 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Advanced and/or metastatic solid tumor
  * Advanced or metastatic non-Hodgkin's lymphoma refractory to standard therapy
* Clinically or radiologically documented disease

  * No tumor marker elevation as only evidence of disease
* No untreated brain or meningeal metastases

  * Treated and stable brain metastases allowed provided they are asymptomatic and do not require steroids

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.25 times upper limit of normal (ULN) OR creatinine clearance ≥ 50 mL/min
* Bilirubin normal
* ALT and AST ≤ 2 times ULN (≤5 times ULN if liver metastases are present)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two effective methods of contraception
* No untreated or uncontrolled hypertension, cardiovascular conditions, or symptomatic cardiac dysfunction
* No active or uncontrolled infections
* No serious illness or medical condition that would preclude study treatment

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior major surgery and recovered
* At least 3 weeks since prior palliative radiotherapy and recovered

  * Low-dose, nonmyelosuppressive radiotherapy may be allowed
* At least 3 weeks since prior chemotherapy for solid tumors and recovered

  * No more than 2 prior cytotoxic chemotherapy regimens for metastatic disease
* At least 4 weeks since prior steroids
* No limitations on prior therapy for patients with non-Hodgkin's lymphoma
* Prior hormonal, immunologic, biologic or signal transduction inhibitor therapy allowed
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-01-30 (Actual); Primary Completion 2010-04-09 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of Aurora kinase inhibitor AT9283 (AT9283) | 1 year
  Doses escalated as described in protocol section 4.3. MTD defined as that dose at which ≥ 2/6 or ≥ 2/3 patients experience DLT (as defined in protocol section 4.4).
Recommended phase II dose of AT9283 | 1 year
  RPTD defined as one dose lower than MTD.
Safety, tolerability, toxicity profile, and dose-limiting toxicity of AT9283 | every 3 weeks
  Adverse events graded using NCI CTCAE V3.0
Pharmacokinetic profile of AT9283 | cycle one only
  PK samples collected on all patients during cycle 1 as described in protocol section 17.2.

SECONDARY OUTCOMES:
Efficacy of AT9283 | every 6 weeks
  All patients with measurable disease were assessed for response using RECIST criteria as described in protocol section 10.

CONTACTS AND LOCATIONS:
Overall Officials: Karen A. Gelmon, MD, Study Chair — British Columbia Cancer Agency; Susan F. Dent, MD, Study Chair — Ottawa Regional Cancer Centre
Locations (2):
- Canada (2):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dent SF, Gelmon KA, Chi KN, Jonker DJ, Wainman N, Capier CA, Chen EX, Lyons JF, Seymour L. NCIC CTG IND.181: phase I study of AT9283 given as a weekly 24 hour infusion in advanced malignancies. Invest New Drugs. 2013 Dec;31(6):1522-9. doi: 10.1007/s10637-013-0018-9. Epub 2013 Sep 27. PMID 24072436